CLINICAL TRIAL: NCT00260949
Title: Functional and Anatomical Results Following Arthroscopic Cuff Repair
Brief Title: Outcome Following Surgery to Repair Rotator Cuff Tears
Status: Terminated | Type: Observational
Why Stopped: As per advice from clinicaltrials.gov, study was mistakenly entered. Since ClinicalTrials.gov is unable to remove the record, they suggested we change the study status. Adjusting the status would eliminate the reporting requirements.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2003534-01H
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear; arthroscopic repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Arthroscopic repair of rotator cuff tear — Patients will undergo arthroscopic shoulder surgery in the standard fashion

SUMMARY:
There are two ways in which surgeons repair rotator cuff tears. An open method involves making an incision (cut) 5-6 inches in length in the skin and repairing the tear with the skin open, while the arthroscopic method involves making small holes in the skin and using a guiding camera and special equipment to repair the tear. This clinical study is being conducted to study the rate of re-tear (one year following surgery) of rotator cuffs that have been repaired using the arthroscopic technique.

DETAILED DESCRIPTION:
While many studies have researched re-tear rate for rotator cuff tears following open repair, to date there have been no studies evaluating re-tear rate following arthroscopic surgery. Arthroscopic rotator cuff repair is less invasive and exposes the patient to fewer risks than open surgery. Once this pilot study is completed the next step will be to compare the rate of re-tear, as assessed via Magnetic Resonance Imaging (MRI) between the two techniques. If the rate of re-tear is lower following arthroscopic surgery this will provide validation for use of the arthroscopic technique. If, however, the rate of re-tear is higher using the arthroscopic technique, then use of this technique is not justified.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of rotator cuff tear which will involve one of the following:1) history of shoulder pain or weakness 2) ability to illicit pain or weakness with one of the following signs: tenderness of the rotator cuff insertion, palpable crepitus of the subacromial bursa or a palpable defect of the cuff insertion, impingement signs and weakness of the rotator cuff musculature 3) radiological evidence of rotator cuff tear from ultrasound, arthrogram or MRI. Failed non-operative treatment. Size of tear of less than 5 cm and involving 2 or fewer tendons

Exclusion Criteria:

* Clinical:1. Tear as defined by significant muscular wasting, inability to actively forward-flex (strength grade 2/5 or worse), positive drop sign or hornblowers 2. Significant tenderness of acromioclavicular or sternoclavicular joints on affected side3. Presence of comorbid shoulder instability or evidence of SLAP lesion4. Previous surgery on affected shoulderRadiological:1. Bony abnormality on standardized series of x-rays consisting of a minimum of an antero-posterior view, lateral “Y” view in the scapular plane, and an axillary view.2. Presence of massive cuff tear on MRI or ultrasound (defined as > 5 cm or greater than 2 tendons torn).Arthroscopic:1. Presence of massive cuff tear as defined above on arthroscopic examination of the joint 2. Presence of comorbid conditions: Bankart lesion, SLAP lesion3. Inability to complete the repair arthroscopically (eg. partial repair by marginal convergence without direct repair to bone)Other:Patients who have any contraindication to MRI (including claustrophobia, intracranial aneurism clip, cardiac pacemaker, middle ear prosthesis, metallic heart valve prosthesis, prior metal fragment in eye (intraocular lens implant) etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be screened by participating surgeons in a fellowship-run outpatient shoulder clinic. Patients who have consented and are scheduled to undergo an arthroscopic rotator cuff repair, and who have a cuff tear size of <5 cm, and involving 2 or fewer tendons, and meet the additional eligibility criteria will be approached to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Rate of re-tear at 1 year | 1 year
  The rate of rotator cuff re-tear will be measured 1-year post-operatively using a Magnetic Resonance Imaging (MRI) Arthrogram.

SECONDARY OUTCOMES:
Functional Status Anatomical integrity | 1 year
  Overall functional status will be assessed by the American Shoulder and Elbow Surgeons (ASES), which is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome. Functional status will also be assessed using The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points. The test is divided into four sub-categories: (1) pain (2) activities of daily living ability; (3) mobility; (4) strength. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Lapner PC, Su Y, Simon D, El-Fatori S, Lopez-Vidriero E. Does the upward migration index predict function and quality of life in arthroscopic rotator cuff repair? Clin Orthop Relat Res. 2010 Nov;468(11):3063-9. doi: 10.1007/s11999-010-1457-7. Epub 2010 Jul 7. PMID 20607465